CLINICAL TRIAL: NCT07380048
Title: Postural Reeducation: Effects On Spinal Posture And Pain In Adolescents Using Digital Screens
Brief Title: Postural Reeducation to Improve Spinal Posture and Pain in Adolescents Who Use Digital Screens
Acronym: POSTURE-SCREEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Ercília Patricia Oliveira Costa, Principal Investigator (PhD Student), University of Vigo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 04-181233
Record Dates: First submitted 2025-12-27; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Musculoskeletal Pain
Keywords: Adolescent; Body Posture; Physical Education; Global Postural Reeducation; Back Pain; Electronic Devices
MeSH Terms: conditions — Musculoskeletal Pain; Back Pain

STUDY DESIGN:
Intervention Model Description: Participants were assigned to two parallel groups: an experimental group receiving a 12-week postural reeducation program and a control group performing the usual Physical Education warm-up. Outcomes were assessed at baseline and post-intervention.
Masking Description: This is an open-label study. Neither participants nor investigators were blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Experimental (Experimental): Participants assigned to the experimental group will receive a 12-week postural reeducation program integrated into Physical Education classes. The program includes strength and mobility exercises for the spine and shoulder girdle and active global stretching postures designed to improve flexibility and postural control. Sessions are delivered twice per week for 15 minutes at the beginning of the class.
  Interventions: Behavioral: Global Postural Reeducation Program
- Arm 2 - Control (No Intervention): Participants assigned to the control group will follow their usual Physical Education classes and standard warm-up routines. They will not receive any specific postural reeducation program or additional structured exercises beyond the regular school curriculum.

INTERVENTIONS:
Behavioral: Global Postural Reeducation Program — Behavioral: Global Postural Reeducation program The intervention consists of a 12-week school-based program integrated into Physical Education classes. Students perform two 15-minute sessions per week including strengthening and mobility exercises for the spine and shoulder girdle, followed by active global stretching postures aimed at improving flexibility and postural control.
  Other Names: Global Postural Reeducation (RPG); Active Global Stretching; School physical education postural program
  Arms: Arm 1 - Experimental

SUMMARY:
This study evaluated whether a postural reeducation program could improve spinal posture and reduce musculoskeletal pain in adolescents who frequently use digital devices. Prolonged screen use is common among students and is often associated with inadequate sitting or standing postures, which may increase back and neck pain.

A total of 187 adolescents participated in the study. Students were assigned to an experimental group or a control group. The experimental group received a 12-week intervention integrated into the warm-up phase of Physical Education classes, while the control group continued with the usual warm-up used in these classes. The experimental group performed two sessions per week, each lasting 15 minutes, at the beginning of the class. Initially, students completed strength and mobility exercises for the spine and shoulder girdle. From the third week onward, active global stretching postures were added to improve flexibility and postural control.

Spinal posture was assessed at baseline and after the intervention using a noninvasive device (SpinalMouse®). Pain and postural habits were evaluated using a validated questionnaire. Adolescents who participated in the postural reeducation program showed improvements in postural alignment and functional mobility, as well as reductions in back and neck pain, compared with the control group.

This study suggests that a brief school-based postural reeducation program may be an effective preventive strategy to promote spinal health and reduce musculoskeletal pain in adolescents.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of a school-based postural reeducation program on spinal posture, functional mobility, and musculoskeletal pain in adolescents enrolled in lower secondary education (middle school level) who frequently use digital devices. Prolonged use of mobile phones, tablets, and other electronic devices is highly prevalent in this population and is associated with inadequate sitting and standing postures, increased thoracic kyphosis, and greater prevalence of neck and back pain. Preventive strategies implemented in school settings may help mitigate these negative musculoskeletal outcomes.

The primary objective of this study is to determine whether a 12-week intervention using a protocol based on strength and mobility exercises, combined with self-postures from the Global Active Stretching method and grounded in the principles of Global Postural Reeducation, integrated into Physical Education (PE) classes, improves spinal alignment and reduces pain perception in adolescents. Secondary objectives include assessing changes in postural habits related to digital device use and spinal mobility.

This is an experimental study with two parallel groups: an experimental group receiving the intervention and a control group continuing the usual PE warm-up. A total of 187 adolescents participated. During the first week, baseline assessment was performed, including spinal posture evaluation and questionnaire administration. The intervention program was then delivered over 12 consecutive weeks.

The intervention was implemented at the beginning of PE classes and consisted of two 15-minute sessions per week. The sessions included strength and mobility exercises for the spine and shoulder girdle based on the protocol proposed by Feng et al. (2018). In addition, active global stretching postures from the Souchard Active Global Stretching (AGS) method were progressively introduced to improve flexibility and postural control.

Spinal morphology in the sagittal plane was assessed at pretest and posttest using the non-invasive SpinalMouse® device. Postural habits and musculoskeletal pain were assessed using the validated Back Pain and Body Posture Evaluation Instrument for Children and Adolescents (BackPEI-CA) questionnaire. All measurements were conducted under standardized conditions to ensure internal validity.

Participation involves minimal risk, limited mainly to temporary muscular discomfort during exercise performance. Potential benefits include improved postural awareness, spinal alignment, mobility, and musculoskeletal health.

This study is expected to contribute evidence supporting the feasibility and effectiveness of brief school-based postural reeducation programs as a low-cost preventive strategy to promote spinal health in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Age between 13 and 15 years.
* Students enrolled in lower secondary education.
* Regular participation in Physical Education classes.
* Absence of recent musculoskeletal injuries.
* Absence of medical conditions limiting physical activity.
* Completion of the baseline questionnaire.
* Written informed consent signed by legal guardians.

Exclusion Criteria:

* Special educational needs preventing participation in the intervention.
* Medical contraindication for participation in Physical Education classes.
* Recent musculoskeletal injury or condition limiting exercise participation.
* Lack of informed consent.
* Failure to complete baseline or post-intervention assessments.

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 187 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Change in sagittal spinal curvature (thoracic kyphosis and lumbar lordosis) | Baseline and 14 weeks (post-intervention)
  Sagittal spinal posture will be assessed using the Spinal Mouse® device at baseline (pre-intervention) and after 14 weeks (post-intervention). Thoracic kyphosis and lumbar lordosis angles will be recorded in degrees (°). The outcome will be expressed as the difference in angular values between baseline and post-intervention and compared between the intervention and control groups.
Change in thoracic and lumbar range of motion | Baseline and 14 weeks (post-intervention)
  Thoracic and lumbar range of motion (ROM) will be assessed using the Spinal Mouse® device at baseline (pre-intervention) and after 14 weeks (post-intervention), during maximum trunk flexion. ROM will be recorded as a global angular value in degrees (°). The outcome will be expressed as the difference in angular values between baseline and post-intervention and compared between the intervention and control groups.

SECONDARY OUTCOMES:
Change in low back pain intensity (BackPEI-CA) | Baseline and 14 weeks (post-intervention)
  Low back pain intensity will be assessed using the Back Pain and Body Posture Evaluation Instrument for Children and Adolescents (BackPEI-CA) at baseline (pre-intervention) and after 14 weeks (post-intervention). Pain intensity will be reported as a questionnaire score. The outcome will be expressed as the change in score between baseline and post-intervention and compared between the intervention and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Águeda Gutiérrez-Sánchez, PhD, Study Director — University of Vigo - Faculty of Education and Sport Sciences; Ercília Oliveira-Costa, PhD Student, Principal Investigator — University of Vigo - Faculty of Education and Sport Sciences
Locations (1):
- Agrupamento de Escolas D. Maria II, Vila Nova de Famalicão, Portugal

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the study involves minors and contains sensitive health-related information. Data will be used exclusively for research purposes within the project team, in accordance with institutional and ethical approvals.